CLINICAL TRIAL: NCT04157621
Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) in Mild to Moderate Parkinson's Disease
Brief Title: taVNS in Mild to Moderate Parkinson's Disease
Acronym: taVNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Vanessa Hinson, Program Director, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00073767
Record Dates: First submitted 2019-09-09; First posted 2019-11-08 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active taVNS (Active Comparator)
  Interventions: Device: Active taVNS
- Sham Stimulation (Sham Comparator)
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Active taVNS — Patients will be masked to transcutaneous stimulation of the auricular branch of the vagus nerve at the tragus
  Arms: Active taVNS
Device: Sham Stimulation — Sham stimulation involves identical perceptual threshold finding and stimulation parameters as active stimulation, with the exception of stimulation target. Sham stimulation will be delivered to the left earlobe, a target believed to have little to no vagal nerve innervation.
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to find out whether a non-invasive form of nerve stimulation called transcutaneous vagus nerve stimulation (taVNS) is safe and effective in people with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-79 y
* Idiopathic Parkinson's Disease Diagnosis
* Disease Stage: Hoehn and Yahr stage 2-3
* Patient requires a minimum of 3 doses of levodopa daily
* Willingness to be videotaped

Exclusion criteria:

* Dementia or Montreal Cognitive Assessment score <24
* Parkinson's Disease psychosis
* Ear trauma
* Facial pain
* Traumatic Brain Injury or clinical history of stroke
* Metal implants above the shoulders
* History of myocardial infarction or arrhythmia, bradycardia
* Active respiratory disorder
* Alcohol or substance use disorders
* History of Deep Brain Stimulation (DBS) or other brain surgery
* Epilepsy
* Pregnancy
* B-Blockers, dopamine blocking agent, antiarrhythmic medication, acetylcholine esterase inhibitor, midodrine, florinef, droxidopa, or anticholinergic drugs

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Hinson, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active taVNS | Sham Stimulation
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active taVNS | Sham Stimulation | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 9 | 11 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor Function Score as Assessed by Modified Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III
Description: The MDS-UPDRS is a rating scale used in research and clinic to rate the severity of Parkinson's Disease. A low score indicates mild disease and a high score more advanced disease. The possible range for MDS-UPDRS Part III is 0-132. Higher scores reflect greater motor disturbance. A decline in score from pre-post would indicate improvement. This outcome observed Part III of UPDRS motor examination.
  Information on cover page:
  The MDS-UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications). Part I has two components: IA concerns a number of behaviors that are assessed by the investigator with all pertinent information from patients and caregivers, and IB is completed by the patient with or without the aid of the caregiver, but independently of the investigator. These sections can, however, be reviewed by the rater to ensure that all questions are answered clea
Time Frame: Baseline (Visit 1) to Day 14 (Visit 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active taVNS | Sham Stimulation
Number analyzed (Participants) | 15 | 15
score on a scale | 0.72 (0.85) | 0.01 (1.02)

2. Secondary Outcome: Change in Cognitive Function Score
Description: Delis-Kaplan Executive Function System (DKEFS) letter fluency is an investigator administered test that assesses verbal fluency. Higher scores indicate more correct responses. A positive value of change means an improvement in fluency. A decrease in score represents decrease in fluency. The minimum score is 0 and there is no maximum score. The raw score is total from letters F, A, and S.
Time Frame: Screening to Day 13 (Visit 9)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active taVNS | Sham Stimulation
Number analyzed (Participants) | 15 | 15
score on a scale | -3.35 (2.58) | 5.12 (2.59)

3. Secondary Outcome: Change in Cognitive Function Score
Description: DKEFS category fluency is an investigator administered test checking into ability to switch between categories presented. There is no upper limit on the D-KEFS measures. There is no lower limit on the D-KEPS measure. Higher scores reflect better verbal fluency. An increase in score from pre-post would indicate improvement. Decrease in value represents decrease in fluency. Raw score is total of Animals + Boys Names.
Time Frame: Screening to Day 13 (Visit 9)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active taVNS | Sham Stimulation
Number analyzed (Participants) | 15 | 15
score on a scale | 1.25 (0.60) | -0.22 (0.83)

4. Secondary Outcome: Change in Cognitive Function Score
Description: Digit span forward is an investigator administered test looking at attention. The possible range for Digit Span Forward is 0-16, same for Digit Span Backward. Higher scores reflect better focused attention and working memory. An increase in score from pre-post would indicate improvement.
Time Frame: Screening to Day 13 (Visit 9)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active taVNS | Sham Stimulation
Number analyzed (Participants) | 15 | 15
score on a scale | 0.19 (0.30) | 0.70 (0.44)

ADVERSE EVENTS:
Time Frame: PI and study coordinator monitored participant safety for 4 weeks
Arm/Group | Active taVNS | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT04157621/Prot_SAP_000.pdf